CLINICAL TRIAL: NCT00900939
Title: Plant-based Dietary Intervention for Treatment of Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acne001
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-fat, vegan diet (Experimental)
  Interventions: Behavioral: Low-fat, vegan diet
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Low-fat, vegan diet — Participants in the intervention group will be asked to follow a low-fat, vegan diet for the full 16 weeks of the study. They will also be guided to favor foods with a low glycemic index. The diet consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products, added oils, and added sugars will be excluded.
  Arms: Low-fat, vegan diet
Behavioral: Control — Participants assigned to the control group will be instructed to follow their usual diets for the full 16 weeks of the study.
  Arms: Control

SUMMARY:
The purpose of this study is to determine if a low-fat, vegan diet affects the number of acne lesions, acne severity, and acne extent.

DETAILED DESCRIPTION:
Acne is the most common skin disorder in the United States. Although many cases are transient, the condition is often chronic, causing self-consciousness and social stigmatization over the short term and physical scars and damaged self-esteem over the long term. Patients and clinicians have frequently attributed acnegenesis to diet; studies of varying quality have been published on the topic since the 1830s. Recently, well-designed, controlled, prospective studies suggest an acnegenic effect of specific dietary factors, including high-glycemic-index foods and dairy products. Limited evidence also suggests an acnegenic effect of foods containing saturated fats. More well-designed, randomized, controlled trials are needed to further establish dietary effects on acne. Based on epidemiologic observations and results of prior clinical trials, we are conducting a pilot study to determine if a low-fat, low-glycemic-index vegan diet affects the number of acne lesions and acne severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female gender
2. Mild, moderate, or severe acne, as indicated by an Evaluator Global Severity Score (EGSS) score of 2, 3, or 4
3. Presence of at least 10 inflammatory or 20 non-inflammatory lesions on the face
4. Presence of acne for at least 3 months (by volunteer's history)
5. Age at least 18 years
6. Ability and willingness to participate in all components of the study
7. Willingness to be assigned randomly to a low-fat, vegan diet or a control group
8. Intention to remain in the Washington DC area for the 16-week study period.

Exclusion Criteria:

1. Change in use or dosage of hormone-based contraceptives in the last 3 months or anticipated change during the study period.
2. Use of depot medoxyprogesterone contraception
3. Use of oral retinoids in the last 6 months
4. Use of high doses of vitamin A in the last 3 weeks (≥ 10,000 IU)
5. Use of oral antibiotics or topical antibacterial or retinoid agents in the last 1 month
6. Presence of more than two nodules or cysts on the face or more than two nodules or cysts on the back and chest.
7. Use of medications known to cause or exacerbate acne including lithium, oral or injected steroids, or medications containing iodides or bromides
8. History of alcohol abuse or dependency followed by any current use
9. Current or unresolved past drug or alcohol abuse
10. Facial hair that would interfere with making acne assessments
11. Pregnancy or breastfeeding (currently or in the past 3 months), or intent to become pregnant in the next 4 months
12. History of severe mental illness within the past 3 years
13. Unstable medical status
14. Current dietary pattern that is low-fat and vegan
15. Anticipated difficulty attending or participating in group sessions
16. Inordinate fear of blood draws
17. Diabetes treated with insulin or any other medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of acne lesions | 16 weeks

SECONDARY OUTCOMES:
Diet acceptability and adherence | 16 weeks
Acne severity and extent | 16 weeks
Quality of life | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Center for Clinical Research, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Spencer EH, Ferdowsian HR, Barnard ND. Diet and acne: a review of the evidence. Int J Dermatol. 2009 Apr;48(4):339-47. doi: 10.1111/j.1365-4632.2009.04002.x. No abstract available. PMID 19335417